CLINICAL TRIAL: NCT02578108
Title: A Prospective Trial of Zero Versus One Diagnostic Genicular Nerve Blocks to Determine Clinical Outcomes After Radiofrequency Ablation for the Treatment of Chronic Painful Knee Osteoarthritis
Brief Title: Diagnostic Genicular Nerve Block Prior to Radiofrequency Ablation for Knee Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Zachary McCormick, MD, Physician, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STU00201206
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis, Knee; Pain; Nerve; Lesion
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Lidocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no diagnostic genicular nerve blocks (Active Comparator): no diagnostic genicular nerve blocks prior to genicular nerve ablation Intervention: genicular nerve radiofrequency ablation
  Interventions: Procedure: genicular nerve radiofrequency ablation
- diagnostic genicular nerve blocks (Active Comparator): Set of diagnostic genicular nerve blocks prior to genicular nerve ablation Intervention: genicular nerve radiofrequency ablation
  Interventions: Procedure: genicular nerve diagnostic block with lidocaine (local anesthetic); Procedure: genicular nerve radiofrequency ablation

INTERVENTIONS:
Procedure: genicular nerve diagnostic block with lidocaine (local anesthetic) — sensory denervation of the knee joint
  Arms: diagnostic genicular nerve blocks
Procedure: genicular nerve radiofrequency ablation — Ablation of the genicular nerves of the knee by radiofrequency energy

SUMMARY:
Chronic painful knee OA is a major cause of disability in older adults. In patients whose symptoms are refractory to conservative management but who do not wish to undergo TKA or, alternatively, are not operative candidates, genicular nerve RFA represents a promising treatment option.

Investigators will determine if patients with chronic painful knee osteoarthritis experience meaningful and long-term improvement in pain, function, and analgesic use, as well as prevention of TKA after RFA of the genicular nerves. Investigators will also determine whether zero versus one set of diagnostic genicular nerve blocks

Answering these questions will help determine if genicular nerve RFA is indeed a worthwhile treatment for chronic painful knee OA. Additionally, this will help determine the optimal diagnostic protocol for patient selection for this procedure, which has implications for improving treatment success rates, preventing unnecessary procedures, and decreasing healthcare cost savings.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the most common conditions and causes of disability in older adults, with an estimated prevalence of symptoms in 20-30% of individuals over 65 years of age. Pain associated with knee OA may have a central nervous system component, but intra-articular chemical pain mediators such as Substance P and Calcitonin-gene related peptide, possible intra-articular ischemic pain due to vasospasm, mechanical compression or irritation of the richly innervated subchondral bone, periosteum, synovium, and joint capsule, as well as peripheral genicular nerve sensitization have largely been implicated.

Knee OA, in general, is treated conservatively with weight loss (when indicated), physical therapy, oral analgesic medications, and intra-articular corticosteroid or hyaluronic acid injections. If this approach fails to provide adequate pain relief and functional restoration, patients may be offered total knee arthroplasty (TKA), if they are surgical candidates. While, TKA is generally a safe procedure, like any major open surgery, it is associated with a risk of serious complications; a large cohort study of 83,756 patients demonstrated the annual incidence of venous thromboembolism (0.6%), myocardial infarction (0.5%), stroke (0.5%), and a 90 day mortality (0.7%) to all be significantly higher than the general population. Furthermore, some patients are not candidates for TKA due to co-morbidities such as morbid obesity or cardiopulmonary disease.

Radiofrequency ablation (RFA) for knee joint denervation represents a promising intervention for patients with chronic painful knee osteoarthritis who have failed conservative management and are either not willing or not eligible for TKA. During RFA a thermal lesion is created by applying radiofrequency energy through an electrode placed at a target structure. RFA has been used to disrupt sensory afferent nociceptive nerve fibers supplying the zygapophyseal (facet) joints of the spine as well as the sacroiliac joint with excellent pain reduction and functional improvement when performed appropriately.

To date, there are only two published studies that have investigated knee joint denervation by RFA for the treatment of chronic painful OA. In a randomized prospective study (n=35), Choi et al. found that genicular nerve RFA resulted in clinically meaningful pain improvement in approximately 60% of patients at 6 month follow-up. Improvement in function was also observed. Bellini and Barbieri report a series of 3 patients with chronic painful knee OA, two of whom who experienced meaningful pain and functional improvement after genicular nerve RFA.

There is no evidence-based algorithm established which provides a means of properly selecting which patients would benefit from genicular nerve RFA. In the study performed by Choi et al., only one set of diagnostic genicular nerve blocks with a threshold of 50% pain relief to be considered a "positive response" was used. In contrast, a well developed literature regarding selection of patients for medial branch RFA for facet-mediated pain indicates that two sets of diagnostic medial branch nerve blocks with a threshold of >80% pain reduction to be considered a "positive response" increased positive predictive value for both meaningful pain and functional outcomes to 80-90%. While the diagnosis of facet-mediated pain can be challenging given the variety of potential pain generators in the spine, diagnostic uncertainly is far less likely when evaluating the knee as a pain generator. In fact, it is unclear that any diagnostic blocks of the genicular nerves are needed given that this increase the potential for complications and healthcare costs compared to proceeding directly to the ablation procedure. It is vital that evidence-based selection criteria are developed for genicular nerve RFA in order to optimize clinical outcomes and minimize healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. All patients ages 30-80 with chronic painful knee osteoarthritis who would undergo treatment by genicular nerve radiofrequency ablation.
2. Knee pain for at least 6 months.
3. Kellgren-Lawrence knee osteoarthritis of 2 or greater.
4. Pain resistant to conventional therapy including NSAIDs, opioids, muscle relaxants, oral steroids, physical therapy, and intra-articular injection therapy.
5. No pain referral beyond the expected distribution for knee osteoarthritis.

Exclusion Criteria:

1. NRS pain score of 4 or more
2. Focal neurologic signs or symptoms.
3. Previous radiofrequency ablation treatment for similar symptoms.
4. Intra-articular knee corticosteroid or hyaluronic acid injection in the past 3 months.
5. Concomitant radicular pain.
6. Previous knee surgery.
7. Patient refusal.
8. Lack of consent.
9. Active systemic or local infections at the site of proposed needle and electrode placement.
10. Coagulopathy or other bleeding disorder, current use of anticoagulants or anti-platelet medications.
11. Allergy to medications being used for injection procedures (contrast, local anesthetic).
12. Inability to read English, communicate with staff, or participate in follow-up.
13. Pregnancy.
14. Pacemaker.
15. Cognitive deficit.
16. Unstable medical or psychiatric illness.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
>50% relief of pain from before to after radiofrequency ablation of the genicular nerves | 6 months
  Outcomes will be compared between those who received a set of diagnostic blocks and those who did not receive a set of diagnostic blocks (arm 1 vs. arm 2)

SECONDARY OUTCOMES:
Mean reduction in morphine equivalent use for knee pain from before to after radiofrequency ablation of the genicular nerves | 6 months
  Outcomes will be compared between those who received a set of diagnostic blocks and those who did not receive a set of diagnostic blocks (arm 1 vs. arm 2)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary McCormick, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States